CLINICAL TRIAL: NCT01874977
Title: Randomized Controlled Trial of a Physical Activity Intervention for RA Fatigue
Brief Title: Trial of a Physical Activity Intervention for RA Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Patti Katz, Professor of Medicine, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CA-0047102
Record Dates: First submitted 2013-06-05; First posted 2013-06-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; fatigue; physical activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pedometer only (Experimental): This group will receive the educational booklet and discussion, plus a pedometer and a diary to record their daily step counts from the pedometer. Participants will be shown how to wear the pedometer, and instructed to wear it from the time they get out of bed in the morning until they go to bed at night, except while showering or bathing. (If any subjects begin a swimming- or cycling-based activity program, we will ask them to remove the pedometer at that time but track the time they are in the water. Step counts will be adjusted to account for this time by adding 150 steps for every minute engaged in swimming and/or cycling.)
  Interventions: Behavioral: Pedometer; Behavioral: Educational materials
- Pedometer + step count goals (Experimental): Pedometer + step goals. This group will receive the educational booklet and discussion, and the pedometer and step diary, plus will be given individualized daily step targets.
  Interventions: Behavioral: Pedometer; Behavioral: Educational materials; Behavioral: Step count goals
- Education materials (Other): Educational materials. This group will receive the educational booklet ("Be Active Your Way: A guide for Adults"; http://www.health.gov/paguidelines/adultguide/default.aspx).and a discussion of simple ways to increase physical activity in daily life based on the booklet, following the baseline assessment. They will receive follow-up contact at the same time points as the intervention groups, although the Week 0 and Week 1 contacts will be by phone instead of in-person and the content of contacts will be different.
  Interventions: Behavioral: Educational materials

INTERVENTIONS:
Behavioral: Pedometer — Will receive the educational booklet and discussion, plus a pedometer and a diary to record their daily step counts from the pedometer.
  Arms: Pedometer + step count goals; Pedometer only
Behavioral: Educational materials — Will receive the educational booklet ("Be Active Your Way: A guide for Adults"; http://www.health.gov/paguidelines/adultguide/default.aspx).and a discussion of simple ways to increase physical activity in daily life based on the booklet, following the baseline assessment.
Behavioral: Step count goals — Will receive the educational booklet and discussion, and the pedometer and step diary, plus will be given individualized daily step targets.
  Arms: Pedometer + step count goals

SUMMARY:
The major goal of this project is to conduct a randomized, controlled trial of the impact of a practical, low cost physical activity intervention on fatigue among persons with rheumatoid arthritis (RA). Fatigue has been identified as a major concern for individuals with RA, and is considered a core outcome measure for RA. Our recent study of the sources of fatigue identified physical inactivity as a primary predictor of fatigue. Studies have examined the impact of exercise interventions on RA outcomes, but most of these interventions have focused on pain or function as outcomes. The few exercise studies examining fatigue suggest that increasing physical activity reduces fatigue, but the interventions have been resource-intensive, requiring specially trained personnel to administer them, highly structured activities, and/or attendance at classes or a specified facility. Each of these components increases the cost and barriers to implementation of an intervention. Pedometers have been shown to be an effective means of increasing physical activity, and could form the basis of a simple means to increase physical activity.

This project will test the effect of a simple pedometer-based intervention, with two incremental degrees of guidance, on increasing physical activity and decreasing fatigue. Three groups (n=40 in each) will be studied: a control group with an educational pamphlet only, a pedometer-only intervention group, and a pedometer group with step targets. Both intervention groups will keep step-count diaries. Groups will be followed over 20 weeks. We expect that (1) the pedometer-only intervention group will increase activity more than the education group, and the group with step-count targets will demonstrate even greater increases in activity; and (2) greater increases in activity will be associated with greater decreases in fatigue. Secondary outcome measures will include depressive symptoms, self-reported sleep quality, and body composition. Our overall goal is to demonstrate an effective, yet simple and low cost, physical activity intervention to decrease fatigue that could be broadly accessible and have the potential for wide implementation.

ELIGIBILITY:
Inclusion Criteria:

* Physicians' diagnosis of RA
* English verbal fluency
* Residence in the greater San Francisco Bay Area
* Score ≥20 on 10-item PROMIS fatigue scale, or at least one item rated "often"
* BMI ≥ 20 kg/m2

Exclusion Criteria:

* Currently engaging in regular exercise
* Non-ambulatory or presence of a condition or comorbid disease that would limit the ability to engage in walking (e.g., foot deformities, lower extremity joint surgery upcoming or in past 6 months, myocardial infarction in past 6 months, stroke, congestive heart failure, severe chronic obstructive pulmonary disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
PROMIS Fatigue scale | change from baseline fatigue score at 20 weeks

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | change from baseline PHQ-9 score at 20 weeks
  depressive symptoms
Pittsburg Sleep Quality Index (PSQI) | Change from baseline PSQI score at 20 weeks
  self-reported sleep quality
Change in weight | Change from baseline weight at 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Katz, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Katz P, Margaretten M, Gregorich S, Trupin L. Physical Activity to Reduce Fatigue in Rheumatoid Arthritis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Jan;70(1):1-10. doi: 10.1002/acr.23230. Epub 2017 Dec 6. PMID 28378441